CLINICAL TRIAL: NCT04406831
Title: The Role of MicroRNA in the Diagnosis, Prognosis and Response to Treatment in Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Nuvance Health (Other)
Responsible Party: Principal Investigator, Richard Frank, Director of Cancer Research, Nuvance Health
Other Study IDs: 15-10
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer Stage III; Pancreatic Cancer Stage IV; Pancreatic Ductal Adenocarcinoma; Pancreatic Neoplasms
Keywords: Pancreas; Cancer; Biomarker
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New Unresectable Pancreatic Cancer: Individuals with biopsy-proven adenocarcinoma of the pancreas, classified as locally advanced or metastatic disease
  Interventions: Procedure: Blood draw
- Control: Healthy individuals without cancer diagnoses to provide reference microRNA
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Individuals in the unresectable pancreatic cancer group will receive monthly blood draws. Individuals in the control group will receive one blood draw

SUMMARY:
Aberrant miRNA production has been linked to a wide range of human cancers and shown to play important roles in their genesis and growth. These miRNA can be detected in the blood and tumors of patients with cancer. The investigators hypothesize that the detection of certain miRNAs present in the blood/serum of patients with pancreatic cancer may be important to the early diagnosis of the disease. Furthermore, the investigators hypothesize that miRNA detection in PC patients will yield prognostic information and help predict the response to treatment.

DETAILED DESCRIPTION:
Specific aims of the study include:

1. To obtain serum samples from patients with newly diagnosed pancreatic cancer at baseline before treatment and monthly throughout treatment.
2. To analyze the miRNA profiles present at each time point.
3. To determine miRNAs that may distinguish pancreatic patients from unaffected individuals. This could be developed into a diagnostic test.
4. To determine miRNAs whose levels correlate with treatment response, both in patients with and without elevations in the serum tumor marker CA 19-9.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy proven adenocarcinoma of the pancreas
* Have initially inoperable disease, classified as either locally advanced or metastatic disease

  * Recurrent disease after a Whipple procedure is allowed
  * Patients who are able to undergo resection after neoadjuvant therapy will continue to be followed after resection
* Have radiographically measurable disease
* Have an ECOG performance status of 2 or less
* Be willing to contribute the required information and specimens
* Provide written signed consent to participate

Exclusion Criteria:

* Having received prior anti-cancer treatments for metastatic pancreatic cancer
* Concurrently receiving systemic therapy for another cancer except androgen deprivation therapy for stable/controlled prostate cancer
* Presence of other active cancer except for: adequately treated local basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for >1 year prior to start of trial. Other adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for > 5 years is allowable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with new diagnoses of unresectable pancreatic cancer, or recurrent pancreatic cancer following a Whipple procedure
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of miRNA profile | Through study completion, up to 5 years
  Analyze the miRNA profiles present at each time point.

SECONDARY OUTCOMES:
PCR miRNA validation | Through study completion, up to 5 years
  Determine miRNAs that may distinguish pancreatic patients from unaffected individuals. This could be developed into a diagnostic test.
miRNA PCR expression | Through study completion, up to 5 years
  Determine miRNAs whose levels correlate with treatment response, both in patients with and without elevations in the serum tumor marker CA 19-9.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Frank, MD, Principal Investigator — Nuvance Health
Locations (1):
- Nuvance Health, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed on an individual basis post submission. Requestors may be required to sign a data access agreement